CLINICAL TRIAL: NCT01186692
Title: Implantation of the Medtronic Melody Transcatheter Pulmonary Valve (TPV) in Patients With Dysfunctional Right Ventricular Outflow Tract (RVOT) Conduits: A Post-Market Approval Study
Brief Title: Melody® Transcatheter Pulmonary Valve Post-Approval Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D03909
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Results first posted 2016-12-26 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Dysfunctional Right Ventricular Outflow Tract (RVOT) Conduit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Melody TPV Implant (Experimental): Melody® Transcatheter Pulmonary Valve implanted into a dysfunctional RVOT Conduit.
  Interventions: Device: Melody® Transcatheter Pulmonary Valve

INTERVENTIONS:
Device: Melody® Transcatheter Pulmonary Valve — Transcatheter Pulmonary Valve replacement Transcatheter valve implantation into a RVOT conduit in patients with complex congenital heart defects where the conduit has become dysfunctional and where the patient needs invasive intervention.
  Other Names: Melody Transcatheter Pulmonary Valve

SUMMARY:
The purpose of this study is to confirm the short-term hemodynamic effectiveness results achieved by real-world providers are equivalent to the historical control established in the IDE study.

ELIGIBILITY:
Inclusion Criteria:

* Existence of a full (circumferential) RVOT conduit that was equal to or greater than 16 mm in diameter when originally implanted
* Dysfunctional RVOT conduits with a clinical indication for intervention (regurgitation ≥ moderate regurgitation, Stenosis: mean RVOT gradient ≥ 35 mmHg)

Exclusion Criteria:

* Implantation in the aortic or mitral position
* Venous anatomy unable to accommodate a 22-fr size introducer sheath
* Obstruction of the central veins
* Clinical or biological signs of infection including active endocarditis
* Unwilling or unable to provide written informed consent or comply with the follow-up requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaqueline Kreutzer, MD, Principal Investigator — Children's Hospital of University of Pittsburgh Medical Center
Locations (10):
- United States (10):
  - Rady Children's Hospital, San Diego, California
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - CS Mott Children's Hospital, University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas, UT Southwestern, Dallas, Texas
  - Primary Children's Medical Center, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Armstrong AK, Berger F, Jones TK, Moore JW, Benson LN, Cheatham JP, Turner DR, Rhodes JF, Vincent JA, Zellers T, Lung TH, Eicken A, McElhinney DB. Association between patient age at implant and outcomes after transcatheter pulmonary valve replacement in the multicenter Melody valve trials. Catheter Cardiovasc Interv. 2019 Oct 1;94(4):607-617. doi: 10.1002/ccd.28454. Epub 2019 Aug 16. PMID 31419019
- [Derived] Armstrong AK, Balzer DT, Cabalka AK, Gray RG, Javois AJ, Moore JW, Rome JJ, Turner DR, Zellers TM, Kreutzer J. One-year follow-up of the Melody transcatheter pulmonary valve multicenter post-approval study. JACC Cardiovasc Interv. 2014 Nov;7(11):1254-62. doi: 10.1016/j.jcin.2014.08.002. Epub 2014 Nov 17. PMID 25459038
- [Derived] McElhinney DB, Benson LN, Eicken A, Kreutzer J, Padera RF, Zahn EM. Infective endocarditis after transcatheter pulmonary valve replacement using the Melody valve: combined results of 3 prospective North American and European studies. Circ Cardiovasc Interv. 2013 Jun;6(3):292-300. doi: 10.1161/CIRCINTERVENTIONS.112.000087. Epub 2013 Jun 4. PMID 23735475

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled: All subjects enrolled (n=131)
Period: Overall Study
Arm/Group | Enrolled
Started | 131
Completed | 99
Not Completed | 32
Not completed — Not Catheterized | 11
Not completed — Futher testing contraindicated implant | 19
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Cohort: All subjects enrolled.
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 131
Age, Continuous [Median (Standard Deviation); unit: years] | 20.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 87
Region of Enrollment [Number; unit: participants]
  United States | 131

OUTCOME MEASURES:

1. Primary Outcome: Acceptable TPV Hemodynamic Function at Six Months After Successful TPV Implantation
Description: Acceptable TPV hemodynamic function at six months after successful TPV implantation is determined as a composite of the following:
  * Mean RVOT gradient is less than or equal to 30 mmHg as measured by CW Doppler, and
  * Severity of pulmonary regurgitation is less than moderate by Doppler echocardiography, and
  * Free from RVOT conduit reoperation or catheter re-intervention at six months after TPV implantation.
  The endpoint is defined as the percentage of subjects with acceptable TPV hemodynamic function at six months after Melody valve implantation.
Time Frame: 6 months
Population: The implanted >24 hours cohort consists of all subjects who had a Melody TPV implanted which remained implanted for greater than 24 hours. Of this population those with evaluable echo data at 6 months post implant were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Implanted >24 Hours Cohort: The implanted >24 hours cohort consists of all subjects who had a Melody TPV implanted which remained implanted for greater than 24 hours.
Arm/Group | Implanted >24 Hours Cohort
Number analyzed (Participants) | 90
percentage of patients | 96.7 [91.6 to 100]

2. Secondary Outcome: Procedural Success
Description: Procedural success is defined as a composite of the following:
  * The TPV is fixated within the desired location, and
  * The RV-PA peak-to-peak gradient measured in the catheterization lab after TPV implantation is less than 35 mmHg, and
  * There is no more than trivial pulmonary regurgitation by angiography
  * The subject is free from explantation of the TPV at 24 hours post-implant
Time Frame: 6 Months
Population: The attempted implant cohort consists of all subjects who underwent catheterization and a Melody TPV implantation was attempted (Melody TPV valve opened).
Measure: Number; unit: percentage of patients
Groups:
- Attempted Implant Cohort: The attempted implant cohort consists of all subjects who underwent catheterization and a Melody TPV implantation was attempted (Melody TPV valve opened).
Arm/Group | Attempted Implant Cohort
Number analyzed (Participants) | 101
percentage of patients | 92.1

3. Secondary Outcome: Serious Procedural Adverse Events
Description: A procedure-related event is defined as an event that is associated with the implant procedure by the chronology or physiology and was caused by the implant procedure (e.g. rupture of the conduit or damage to an intra-cardiac or intravascular structure by the delivery system).
Time Frame: 6 Months
Population: The catheterized cohort consists of all subjects who underwent catheterization for possible implantation of the Melody TPV.
Measure: Number; unit: percentage of patients
Groups:
- Catheterized Cohort: The catheterized cohort consists of all subjects who underwent catheterization for possible implantation of the Melody TPV.
Arm/Group | Catheterized Cohort
Number analyzed (Participants) | 120
percentage of patients | 19.2

4. Secondary Outcome: Serious Device-related Adverse Events
Description: A device-related event is defined as an event that is associated with the TPV by the chronology or physiology and was caused by the the TPV (e.g. embolization of the TPV and any adverse events which follow).
Time Frame: 6 months
Population: The implanted cohort consists of all subjects who underwent catheterization and a Melody TPV was implanted.
Measure: Number; unit: percentage of patients
Groups:
- Implanted Cohort: The implanted cohort consists of all subjects who underwent catheterization and a Melody TPV was implanted.
Arm/Group | Implanted Cohort
Number analyzed (Participants) | 100
percentage of patients | 11.0

5. Secondary Outcome: Changes in NYHA Functional Classification
Description: Change in NYHA functional class from pre-implant to 6 month post-implant
Time Frame: 6 Months
Population: The implanted >24 hours cohort consists of all subjects who had a Melody TPV implanted which remained implanted for greater than 24 hours. Of this population those with evaluable paired NYHA data were included in the analysis.
Measure: Number; unit: participants
Groups:
- Implanted > 24 Hours Cohort: The implanted >24 hours cohort consists of all subjects who had a Melody TPV implanted which remained implanted for greater than 24 hours.
Arm/Group | Implanted > 24 Hours Cohort
Number analyzed (Participants) | 99
participants
  Changes in NYHA Functional Classification | 93
  Improved | 51
  No Change | 39
  Worsened | 3

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Catheterized Cohort
Serious Adverse Events (participants affected / at risk) | 52/120
Other Adverse Events (participants affected / at risk) | 31/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheterized Cohort (N=120)
Anaemias NEC (Blood and lymphatic system disorders) | 1 (1)
Haematological disorders (Blood and lymphatic system disorders) | 1 (2)
Cardiac disorders NEC (Cardiac disorders) | 1 (1)
Coronary artery disorders NEC (Cardiac disorders) | 1 (2)
Pulmonary valvular disorders (Cardiac disorders) | 3 (3)
Rate and rhythm disorders NEC (Cardiac disorders) | 1 (1)
Supraventricular arrhythmias (Cardiac disorders) | 1 (1)
Ventricular arrhythmias and cardiac arrest (Cardiac disorders) | 2 (9)
Gastrointestinal disorders NEC (Gastrointestinal disorders) | 2 (2)
Nausea and vomiting symptoms (Gastrointestinal disorders) | 1 (1)
diarrhoea (excl infective) (Gastrointestinal disorders) | 1 (1)
Device issues NEC (General disorders) | 1 (1)
Device physical property and chemical issues (General disorders) | 9 (10)
Febrile disorders (General disorders) | 2 (3)
Therapeutic and nontherapeutic responses (General disorders) | 4 (9)
Cardiac infections (Infections and infestations) | 3 (5)
Lower respiratory tract and lung infections (Infections and infestations) | 1 (1)
Sepsis, bacteraemia, viraemia and fungaemia NEC (Infections and infestations) | 1 (2)
Cardiac and vascular procedural complications (Injury, poisoning and procedural complications) | 1 (1)
Non-site specific procedural complications (Injury, poisoning and procedural complications) | 4 (5)
Nervous system disorders NEC (Nervous system disorders) | 1 (3)
Neurological signs and symptoms NEC (Nervous system disorders) | 1 (2)
Pneumothorax and pleural effusions NEC (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Pulmonary thrombotic and embolic conditions (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory tract disorders NEC (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Non-site specific embolism and thrombosis (Vascular disorders) | 2 (5)
Vascular injuries NEC (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheterized Cohort (N=120)
Pain and discomfort NEC (General disorders) | 8 (9)
Therapeutic and nontherapeutic responses (General disorders) | 8 (13)
Infections NEC (Infections and infestations) | 7 (8)
Non-site specific procedural complications (Injury, poisoning and procedural complications) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A publication committee is in place for this study.